CLINICAL TRIAL: NCT05371717
Title: Management of Dental Erosion in Patients With Gastroesophageal Reflux Disease With Biomimetic Hydroxyapatite Toothpaste
Brief Title: Domiciliary Management of Dental Erosion in Patients With GERD With Biomimetic Hydroxyapatite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-GASTRO
Record Dates: First submitted 2022-05-03; First posted 2022-05-12 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Gastro Esophageal Reflux; Dental Erosion
Keywords: biomimetic hydroxyapatite; remineralization
MeSH Terms: conditions — Gastroesophageal Reflux; Tooth Erosion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial Group (Experimental): Domiciliary use of Biorepair Total Protection + Biorepair Shock Treatment application
  Interventions: Other: Domiciliary use of Biorepair Total Protection + Biorepair Shock Treatment
- Control group (Active Comparator): Domiciliary use of Biorepair Total Protection
  Interventions: Other: Biorepair Total Protection

INTERVENTIONS:
Other: Domiciliary use of Biorepair Total Protection + Biorepair Shock Treatment — Domiciliary use of Biorepair Total Protection twice a day for oral hygiene + Biorepair Shock Treatment application for 10 min once a day.
  Arms: Trial Group
Other: Biorepair Total Protection — Domiciliary use of Biorepair Total Protection twice a day for oral hygiene + Biorepair Shock Treatment application for 10 min once a day.
  Arms: Control group

SUMMARY:
The aim of the present study is to evaluate dental erosion in patients with gastroesophageal reflux disease (GERD).

Patients consenting to participate to the study will undergo periodontal evaluation at the baseline. Then, professional dental hygiene will be performed. Patients will be randomly assigned to:

* Trial group: home oral hygiene with Biorepair Total Protection + Biorepair Shock Treatment twice a day
* Control group: home oral hygiene with Biorepair Total Protection Patients will be evaluated after 1, 3, 6, 9 and 12 months from baseline.

DETAILED DESCRIPTION:
The aim of the present study is to evaluate dental erosion in patients with gastroesophageal reflux disease (GERD).

Patients consenting to participate to the study will undergo periodontal evaluation at the baseline. Then, professional dental hygiene will be performed. Patients will be randomly assigned to:

* Trial group: home oral hygiene with Biorepair Total Protection + Biorepair Shock Treatment twice a day
* Control group: home oral hygiene with Biorepair Total Protection Patients will be evaluated after 1, 3, 6, 9 and 12 months from baseline.

ELIGIBILITY:
Inclusion Criteria:

* patients with dental erosion
* no proton pumps before pH examination

Exclusion Criteria:

* no dental erosion
* neurological and psychiatric diseases;
* pregnant and/or breastfeeding women;
* patients with poor compliance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Change of BEWE (Basic Erosive Wear Examination) | Study begin, 1, 3, 6, 9 and 12 months after the baseline
  Scoring criteria (Barlet et al., 2008):
  * 0: no erosive tooth wear;
  * 1: initial loss of surface texture;
  * 2: distinct defect, hard tissue loss < 50% of the surface area;
  * 3: hard tissue loss ≥ 50% of the surface area.
  IntactTooth smartphone application will be used to calculate this index.
Change in Schiff Air Index - Dental sensitivity test | Study begin, 1, 3, 6, 9 and 12 months after the baseline
  Scoring criteria:
  0: the subject did not respond to air blasting;
  1. the subject responded to air blasting;
  2. the subject responded to air blasting and requested discontinuation;
  3. the subject responded to air blasting, requested discontinuation and considered the stimulus to be painful.
Change in Plaque Index (PI% - O' Leary Index) | Study begin, 1, 3, 6, 9 and 12 months after the baseline
  Evaluation of the presence of plaque on the 4 surfaces of teeth on the total amount of dental surfaces.
  Formula = n ° sites with plaque / total n ° of dental surfaces x100
Change in Bleeding Score (BS - Mombelli et al.) | Study begin, 1, 3, 6, 9 and 12 months after the baseline
  Scoring criteria:
  0: no bleeding
  1. isolated visible spots
  2. blood forms a confluent red line on the mucosal margin
  3. profuse and copious bleeding
Laryngopharyngeal pH monitoring | Study begin, 1, 3, 6, 9 and 12 months after the baseline
  Data was collected wirelessly for 24 hours and then analysed. Length, severity and number of reflux episodes were calculated. The RYAN score was used to evaluate for laryngopharyngeal acid reflux and was calculated for both the upright and supine positions. A RYAN score >9.4 in the upright position or >6.8 in the supine position was considered positive. Patients with a positive RYAN score in either the upright or supine positions were considered positive for laryngopharyngeal acid reflux.
Erosion risk level | Study begin, 1, 3, 6, 9 and 12 months after the baseline
  For each sextant, the highest BEWE value will be chosen. A mean of all the sextant values will be performed to calculate erosion risk level.
  IntactTooth smartphone application will be used to calculate this index.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, MS, Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator.